CLINICAL TRIAL: NCT02005718
Title: Impact of Cholecalciferol on Endothelial Fucntion and Blood Biomarkers in Patients With Chronic Kidney Disease
Brief Title: Impact of Vitamin D on Endothelial Function and Blood Biomarkers Including CD28 Null Cells in CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090129
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: CKd Patients With Stage 3 and 4
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D (Experimental): Cholecalciferol 300,000 twice
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol

SUMMARY:
Vitamin D deficiency is common in CKD and assciated with CV complications. Endothelial dysfucntion is common in CKD and is a harbinger of atherosclerosis. The study investigated the impact of Vitamin D on endothelial fucntion and blood biomarkers in CKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD 3-4 Age 18-80

Exclusion Criteria:

* Recent MI, CVA, malignancy active infection active inflammation High calcium already on Viatmin D therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | 16 weeks

SECONDARY OUTCOMES:
CD28 null cell frequency | 16 weeks
Blood biomarkers of endothelial function and inflammation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Banerjee, Principal Investigator — St Georges

REFERENCES:
- [Derived] Chitalia N, Ismail T, Tooth L, Boa F, Hampson G, Goldsmith D, Kaski JC, Banerjee D. Impact of vitamin D supplementation on arterial vasomotion, stiffness and endothelial biomarkers in chronic kidney disease patients. PLoS One. 2014 Mar 19;9(3):e91363. doi: 10.1371/journal.pone.0091363. eCollection 2014. PMID 24646518